CLINICAL TRIAL: NCT05892419
Title: Electrophysiological Signatures of Distinct Working Memory Subprocesses That Predict Long-term Memory Success
Acronym: WMLTM
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB15-1290
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Memory; EEG

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — There is no intervention

SUMMARY:
Healthy young adults will view pictures of items while the investigators record electroencephalogram (EEG) brain activity. Then, the investigators will ask the participants to report which items the participants remember seeing. The investigators will examine how the measured brain activity relates to which pictures the participants remember.

DETAILED DESCRIPTION:
Electrophysiological signatures track distinct subprocesses of working memory, including the number of items and the spatial locations of those items. By identifying how these subprocesses predict long-term memory success in healthy young adults, this project should lead to an intricate understanding of the relationship between working memory and long-term memory. This study will investigate when and how long-term memory failures arise, by using sophisticated machine learning analyses of neural data. Moreover, this study will test the extent to which the investigators can track working memory processes in real time and how the investigators can leverage that information to improve long-term memory success. This will inform basic theories of the relationship between working memory and long-term memory and motivate future applications.

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected to normal vision

Exclusion Criteria:

* non-fluent in English

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Healthy young adults
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Memory performance | This task is performed multiple time within the experimental session, which in total lasts around 3 hours.
  To measure recognition memory performance, participants will view pictures and respond as to whether they remember previously seeing these items. Participants will be shown both old and new items. In the long-term memory phase, they will report their confidence at having seen each image using a four point rating scale, ranging from being confident the item is new (i.e., not previously seen) to being confident the item is old (i.e., previously seen).

CONTACTS AND LOCATIONS:
Overall Officials: Megan deBettencourt, Principal Investigator — University of Chicago; Ed Vogel, Principal Investigator — University of Chicago; Ed Awh, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will post de-identified data online on scientific repositories including the Open Science Framework (online), zenodo or github, so that anonymized data will be made available to outside researchers. Shared data will include, at a minimum, csv or text files that summarize participants performance. Any computer scripts or stimuli used for task development also will be shared.
Supporting Information: Analytic Code
Time Frame: After publication, in perpetuity
Access Criteria: The code and data will be freely available through online repositories.